CLINICAL TRIAL: NCT05839782
Title: Long Term Results in Redo Mitral Valve Surgery After Mitral Valve Repair
Status: Completed | Type: Observational
Sponsor: Michele De Bonis (Other)
Responsible Party: Sponsor-Investigator, Michele De Bonis, Chief of Cardiac Surgery of Advanced and Research Therapies, Ospedale San Raffaele
Organization: Ospedale San Raffaele (Other)
Other Study IDs: LORESAR
Record Dates: First submitted 2023-01-27; First posted 2023-05-03 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Degenerative Mitral Valve Disease
MeSH Terms: interventions — phospholemman

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Re-PLM: Patient in which a new mitral valve repair is performed to treat failed mitral valve repair
  Interventions: Procedure: Mitral valve repair (PLM)
- Re-SVM: Patient in which a mitral valve replacement is performed to treat failed mitral valve repair
  Interventions: Procedure: Mitral valve replacement

INTERVENTIONS:
Procedure: Mitral valve repair (PLM) — A mitral valve plasty is performed to treat mitral regurgitation
  Groups: Re-PLM
Procedure: Mitral valve replacement — A mitral valve replacement with a prosthesis is performed to treat mitral regurgitation
  Groups: Re-SVM

SUMMARY:
The current gold standard for severe mitral regurgitation is mitral valve plasty (PLM). The surgery allows the repair of the mitral valve, therefore without the need for mitral valve replacement (SVM), which involves the implantation of a biological prosthesis or a mechanical prosthesis.

However, PLM has a rate of failure, between 1-4% per year in degenerative mitral pathologies. As a result, patients with PLM failure and severe residual regurgitation are increasingly presenting in recent years.

Generally these patients are re-operated to replace the mitral valve. Our aim is to investigate the differences in re-operation involving mitral valve replacement or re-repair in patients who underwent mitral valve re-operation (re-repair or replacement) in our center between 2003 and 2017.

ELIGIBILITY:
Inclusion Criteria:

* adult patients
* failure of previous mitral valve repair which needed a new surgical treatment
* group Re-PLM: patients reoperated with a new mitral valve repair
* group Re-SVM: patients reoperated with a mitral valve replacement

Exclusion Criteria:

* urgent/emergent procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a failure of mitral valve repair. The patients are divided in 2 groups depending on type of reintervention: a new mitral valve repair (PLM) or mitral valve replacement (SVM)
Sampling Method: Non-Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2019-10-05 (Actual); Primary Completion 2019-10-15 (Actual); Study Completion 2019-10-15 (Actual)

PRIMARY OUTCOMES:
Survival after reintervention | through study completion, a minimum of 2 years
  Time of survival after reintervention for failed mitral valve repair

SECONDARY OUTCOMES:
Risk factors for reintervention | through study completion, a minimum of 2 years
  Identification of predictors of reintervention after mitral valve repair

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Ospedale San Raffaele - Cardiac Surgery Department, Milan, Italy

IPD SHARING:
Plan to Share IPD: No